CLINICAL TRIAL: NCT06298097
Title: Brain Connectivity Measured With High-density Electroencephalography: a Novel Neurodiagnostic Tool for Stroke
Brief Title: Brain Connectivity Measured With High-density Electroencephalography
Acronym: NEUROCONN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019.11
Record Dates: First submitted 2024-02-13; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: high-density electroencephalography; brain connectivity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stroke patients (Other): Resting-state networks obtained through electroencephalography will be analyzed in a group of stroke patients.
  Interventions: Device: Connectivity measures
- healthy participants (Other): Resting-state networks obtained through electroencephalography will be analyzed in a group of healthy participants.
  Interventions: Device: Connectivity measures

INTERVENTIONS:
Device: Connectivity measures — Electroencephalography connectivity measures will be collected and compared in both stroke patients and healthy participants. Connectivity measures will be extracted using these devices: high-density electroencephalography (using either a 128-channel or a 256-channel system) and magnetic resonance imaging.

SUMMARY:
Emerging scientific results show that disrupted functional connectivity in stroke can explain behavioral impairments and predict their recovery over time. However, no technique is yet available for widespread use in clinics to examine how neural synchronization in brain networks is altered in stroke patients. This is crucial to determine favorable prognostic factors and to define individualized rehabilitation protocols. Importantly, the investigators have successfully used high-density electroencephalography (hdEEG) in healthy individuals to measure neural synchronization in brain networks. In this project, the investigators will develop methods and tools based on hdEEG for assessing functional connectivity in stroke patients. These methods and tools will be employed to examine how neural changes occurring after brain lesions explain behavioral impairments. The project will open the way for the use of hdEEG at the patient's bedside, as a neurodiagnostic tool for stroke as well as other brain disorders.

ELIGIBILITY:
In this study 125 stroke patients and 45 healthy participants will be recruited at the Institute for Research and Healthcare with a Scientific Character (IRCCS) San Camillo hospital.

Inclusion Criteria (patients):

* right or left hemisphere damage
* unilateral stroke
* compliance with magnetic resonance imaging (e.g., no claustrophobia)

Inclusion Criteria (healthy participants):

• compliance with magnetic resonance imaging (e.g., no claustrophobia)

Exclusion Criteria (both patients and healthy participants):

• no comorbidities with psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
High-density electroencephalography measurements (work package 1, 2, and 3) | Immediately after the recruiting
  High-density electroencephalography measurements, specifically focusing on resting state networks, will be performed using either a 128-channel or a 256-channel system
High-density electroencephalography measurements (work package 1, 2, and 3) | 1 month after the recruiting
  High-density electroencephalography measurements, specifically focusing on resting state networks, will be performed using either a 128-channel or a 256-channel system
High-density electroencephalography measurements (work package 1, 2, and 3) | 2 months after the recruiting
  High-density electroencephalography measurements, specifically focusing on resting state networks, will be performed using either a 128-channel or a 256-channel system
High-density electroencephalography measurements (work package 1, 2, and 3) | 4 months after the recruiting
  High-density electroencephalography measurements, specifically focusing on resting state networks, will be performed using either a 128-channel or a 256-channel system
High-density electroencephalography measurements (work package 1, 2, and 3) | 6 months after the recruiting
  High-density electroencephalography measurements, specifically focusing on resting state networks, will be performed using either a 128-channel or a 256-channel system
Magnetic Resonance Imaging measurement (work package 1, 2, and 3) | Immediately after the recruiting
  Magnetic Resonance Imaging will be conducted using a 3 Tesla scanner. Specifically, T1-weighted Magnetic Resonance Imaging measure will be collected
Magnetic Resonance Imaging measurement (work package 1, 2, and 3) | 1 month after the recruiting
  Magnetic Resonance Imaging will be conducted using a 3 Tesla scanner. Specifically, T1-weighted Magnetic Resonance Imaging measure will be collected
Magnetic Resonance Imaging measurement (work package 1, 2, and 3) | 2 months after the recruiting
  Magnetic Resonance Imaging will be conducted using a 3 Tesla scanner. Specifically, T1-weighted Magnetic Resonance Imaging measure will be collected
Magnetic Resonance Imaging measurement (work package 1, 2, and 3) | 4 months after the recruiting
  Magnetic Resonance Imaging will be conducted using a 3 Tesla scanner. Specifically, T1-weighted Magnetic Resonance Imaging measure will be collected
Magnetic Resonance Imaging measurement (work package 1, 2, and 3) | 6 months after the recruiting
  Magnetic Resonance Imaging will be conducted using a 3 Tesla scanner. Specifically, T1-weighted Magnetic Resonance Imaging measure will be collected

SECONDARY OUTCOMES:
Muscle strength measurement (work package 3) | Immediately after the recruiting
  Muscle strength will be measured in the patients by using the Medical Research Council Score
Muscle strength measurement (work package 3) | 1 month after the recruiting
  Muscle strength will be measured in the patients by using the Medical Research Council Score
Muscle strength measurement (work package 3) | 2 months after the recruiting
  Muscle strength will be measured in the patients by using the Medical Research Council Score
Muscle strength measurement (work package 3) | 4 months after the recruiting
  Muscle strength will be measured in the patients by using the Medical Research Council Score
Muscle strength measurement (work package 3) | 6 months after the recruiting
  Muscle strength will be measured in the patients by using the Medical Research Council Score
Sensorimotor impairment measurement (work package 3) | Immediately after the recruiting
  Sensorimotor impairment will be measured in the patients by using the Upper Extremity Fugl-Meyer index
Sensorimotor impairment measurement (work package 3) | 1 month after the recruiting
  Sensorimotor impairment will be measured in the patients by using the Upper Extremity Fugl-Meyer index
Sensorimotor impairment measurement (work package 3) | 2 months after the recruiting
  Sensorimotor impairment will be measured in the patients by using the Upper Extremity Fugl-Meyer index
Sensorimotor impairment measurement (work package 3) | 4 months after the recruiting
  Sensorimotor impairment will be measured in the patients by using the Upper Extremity Fugl-Meyer index
Sensorimotor impairment measurement (work package 3) | 6 months after the recruiting
  Sensorimotor impairment will be measured in the patients by using the Upper Extremity Fugl-Meyer index
Spasticity measurement (work package 3) | Immediately after the recruiting
  Spasticity will be measured in the patients by using the Modified Ashworth Score
Spasticity measurement (work package 3) | 1 month after the recruiting
  Spasticity will be measured in the patients by using the Modified Ashworth Score
Spasticity measurement (work package 3) | 2 months after the recruiting
  Spasticity will be measured in the patients by using the Modified Ashworth Score
Spasticity measurement (work package 3) | 4 months after the recruiting
  Spasticity will be measured in the patients by using the Modified Ashworth Score
Spasticity measurement (work package 3) | 6 months after the recruiting
  Spasticity will be measured in the patients by using the Modified Ashworth Score
Funtional skills measurement (work package 3). | Immediately after the recruiting
  Functional skills will be measured in the patients by using the Functional Independence Measure index. Six domains of function are evaluated: self-care, sphincter control, transfers, locomotion, communication, and social cognition. Self-care activities include dressing, eating, grooming, and bathing.
Funtional skills measurement (work package 3). | 1 month after the recruiting
  Functional skills will be measured in the patients by using the Functional Independence Measure index. Six domains of function are evaluated: self-care, sphincter control, transfers, locomotion, communication, and social cognition. Self-care activities include dressing, eating, grooming, and bathing.
Funtional skills measurement (work package 3). | 2 months after the recruiting
  Functional skills will be measured in the patients by using the Functional Independence Measure index. Six domains of function are evaluated: self-care, sphincter control, transfers, locomotion, communication, and social cognition. Self-care activities include dressing, eating, grooming, and bathing.
Funtional skills measurement (work package 3). | 4 months after the recruiting
  Functional skills will be measured in the patients by using the Functional Independence Measure index. Six domains of function are evaluated: self-care, sphincter control, transfers, locomotion, communication, and social cognition. Self-care activities include dressing, eating, grooming, and bathing.
Funtional skills measurement (work package 3). | 6 months after the recruiting
  Functional skills will be measured in the patients by using the Functional Independence Measure index. Six domains of function are evaluated: self-care, sphincter control, transfers, locomotion, communication, and social cognition. Self-care activities include dressing, eating, grooming, and bathing.
Activities of daily living measurement (work package 3) | Immediately after the recruiting
  Activities of daily living will be measured in the patients by the Barthel Index
Activities of daily living measurement (work package 3) | 1 month after the recruiting
  Activities of daily living will be measured in the patients by the Barthel Index
Activities of daily living measurement (work package 3) | 2 months after the recruiting
  Activities of daily living will be measured in the patients by the Barthel Index
Activities of daily living measurement (work package 3) | 4 months after the recruiting
  Activities of daily living will be measured in the patients by the Barthel Index
Activities of daily living measurement (work package 3) | 6 months after the recruiting
  Activities of daily living will be measured in the patients by the Barthel Index
Pain measurement (work package 3) | Immediately after the recruiting
  Pain level will be measured in the patients by the Visual Analog Scale for Pain
Pain measurement (work package 3) | 1 month after the recruiting
  Pain level will be measured in the patients by the Visual Analog Scale for Pain
Pain measurement (work package 3) | 2 months after the recruiting
  Pain level will be measured in the patients by the Visual Analog Scale for Pain
Pain measurement (work package 3) | 4 months after the recruiting
  Pain level will be measured in the patients by the Visual Analog Scale for Pain
Pain measurement (work package 3) | 6 months after the recruiting
  Pain level will be measured in the patients by the Visual Analog Scale for Pain
Cognitive performance measurements (work package 3) | Immediately after the recruiting
  Cognitive functions will be measured in the patients by using the Oxford Cognitive Screen
Cognitive performance measurements (work package 3) | 1 month after the recruiting
  Cognitive functions will be measured in the patients by using the Oxford Cognitive Screen
Cognitive performance measurements (work package 3) | 2 months after the recruiting
  Cognitive functions will be measured in the patients by using the Oxford Cognitive Screen
Cognitive performance measurements (work package 3) | 4 months after the recruiting
  Cognitive functions will be measured in the patients by using the Oxford Cognitive Screen
Cognitive performance measurements (work package 3) | 6 months after the recruiting
  Cognitive functions will be measured in the patients by using the Oxford Cognitive Screen

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Camillo Hospital, Venice, Italy

IPD SHARING:
Plan to Share IPD: No